CLINICAL TRIAL: NCT02879669
Title: A Randomised Phase II Open-label Study With a Phase Ib Safety lead-in Cohort of ONCOS-102, an Immune-priming GM-CSF Coding Oncolytic Adenovirus, and Pemetrexed/Cisplatin in Patients With Unresectable Malignant Pleural Mesothelioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targovax Oy (Industry)
Collaborators: Theradex (Industry)
Responsible Party: Sponsor
Organization: Targovax ASA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCOS C719; 2015-005143-13 (EudraCT Number)
Record Dates: First submitted 2016-07-13; First posted 2016-08-26 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: To Determine Safety, Tolerability and Efficacy of ONCOS-102 in Combination With Chemotherapy
MeSH Terms: interventions — Pemetrexed; Cisplatin; Carboplatin; Cyclophosphamide

ARMS (2):
- ONCOS-102+cyclophosphamide+pemetrexed/cisplatin (carboplatin) (Experimental): ONCOS-102 will be administered in a priming cycle (Cycle 1) comprising injections on Days 1, 4, 8 and 36, followed by two treatment cycles at intervals of 6 weeks (Cycle 2, Day 78 and Cycle 3, Day 120). Pre-treatment with an i.v. bolus of cyclophosphamide (CPO) will be given 1 to 3 days before the first administration of ONCOS-102 (Cycle 1, Day 1) and before administration of Cycle 2 of ONCOS-102 (Day 78). Patients will also receive pemetrexed/cisplatin (carboplatin) in 21-day cycles starting on Day 22 and continuing as applicable during the study period of 6 cycles of pemetrexed/cisplatin (carboplatin) in combination with ONCOS-102.
  Interventions: Biological: ONCOS-102; Drug: Pemetrexed/cisplatin (carboplatin); Drug: Cyclophosphamide
- Pemetrexed/cisplatin (carboplatin) (Active Comparator): Patients will be treated with pemetrexed/cisplatin (carboplatin) in 21-day cycles starting on Day 1, and continuing as applicable during the study period of 6 cycles of chemotherapy. Patients will be monitored regularly for immunological assessment (PBMCs) including Month 9 and Month 12 (i.e., after the end of study visit), and will be followed up for survival every 3 months until end of life.
  Interventions: Drug: Pemetrexed/cisplatin (carboplatin)

INTERVENTIONS:
Biological: ONCOS-102
  Arms: ONCOS-102+cyclophosphamide+pemetrexed/cisplatin (carboplatin)
Drug: Pemetrexed/cisplatin (carboplatin)
Drug: Cyclophosphamide
  Arms: ONCOS-102+cyclophosphamide+pemetrexed/cisplatin (carboplatin)

SUMMARY:
The trial is an open-label, parallel group, multicentre trial that will recruit a total of 30 patients with malignant pleural mesothelioma. The trial will be conducted in 2 phases: a non-randomised safety phase and a randomised phase. The safety phase will consist of a lead-in cohort of 6 patients treated with ONCOS 102 and pemetrexed/cisplatin. The randomised phase will not commence until the DSMB has deemed the safety lead-in data appropriate for continuation. A total of 24 patients will be included in the randomised phase; 14 patients will be randomised to receive ONCOS 102 and pemetrexed/cisplatin, and 10 patients will receive pemetrexed/cisplatin alone. If cisplatin is seen to be too toxic after one or more cycles, the patient may change to carboplatin during the study. Furthermore, if treatment with cisplatin is deemed to be too toxic by the investigator due to age, presence of neurological toxicities or other relevant medical conditions, carboplatin can be administered from start of study. The trial's main objectives are determination of safety, immune activation, clinical response and the correlation between clinical outcome and the immunological data.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male or female, ≥18 years of age.
* Histologically confirmed unresectable (advanced) malignant pleural mesothelioma in patients who are not candidates for curative surgery and for whom therapy with pemetrexed in combination with cisplatin or carboplatin is considered appropriate. This include:

  * patients who are naïve to chemotherapy,
  * and those who have already received pemetrexed in combination with cisplatin or carboplatin to which their tumour initially responded, but they have relapsed after at least 6 months.

The patient may be evaluated by a multidisciplinary consultation (according to hospital procedure), however the final decision about the inclusion of a patient is made by the principal investigator.

* Measurable disease according to Response Evaluation in Solid Tumour (RECIST 1.1).
* Tumour must be accessible to intratumoural (i.t.) injections and to tumour core needle biopsy or thoracoscopy for tissue sampling and immunohistochemistry analysis.
* The patients must be eligible to receive the study specific chemotherapies, including cyclophosphamide, according to the SPCs and local practice.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance score 0 to 1.
* Acceptable liver, renal, and haematological functions.
* All women of childbearing potential must have a negative urine or serum pregnancy test at screening and all patients must agree to use barrier contraception (i.e. condom) during study treatment and for 2 months after the last virus treatment, 6 months after the last dose of pemetrexed/cisplatin/carboplatin and 12 months after the dose of cyclophosphamide.

Exclusion Criteria:

* Receipt of oncolytic virus treatment, or vaccination with a vaccine containing live virus within 4 weeks before Day 1.
* Use of significant immunosuppressive medication, including high dose corticosteroid (defined as the equivalent of >10 mg/day prednisone) within 4 weeks before Day 1.
* Patients who participated in a study with an investigational drug or device within 4 weeks prior to Day 1.
* Active bacterial, viral, or fungal infections, requiring systemic therapy.
* Severe arrhythmia, heart failure, previous cardiac infarction, or acute inflammatory heart disease.
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient, if included in this study.
* Known infection with HIV, hepatitis B, or hepatitis C.
* Known brain metastases.
* History of organ transplant.
* Females who are pregnant or breast feeding.
* Unwillingness or inability to comply with the study protocol for any reason.
* Patients with pre-existing hearing loss or neuropathy that may worsen due to potential neurotoxicity from cisplatin.
* Patients with a history of hypersensitivity to cisplatin or carboplatin or pemetrexed or cyclophosphamide (or any of its metabolites).
* Patients who are taking phenytoin for prophylactic use.
* History of malignant tumour, unless the patient has been without evidence of disease for at least 3 years, or the tumour was a non-melanoma skin tumour, cervical carcinoma in situ, or prostatic carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06; Primary Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with any (Serious and Non-Serious) Adverse Event measured to assess safety and tolerability | 6 months

SECONDARY OUTCOMES:
To determine and compare tumour-specific immunological activation in the peripheral blood in the experimental group and the control group. Number of patients in the respective arms with induction of Tumor specific CD8+ T Cells in PBMC | 6 months
To determine and compare immunological activation in tumour mass in the experimental group and the control Group. Number of patients in the respective arms with infiltration of CD8+ T Cells into tumours | 6 months
To determine and compare overall response rate in the experimental group and the control group by number of patients with PD, SD, PR and CR in the respective arms | 6 months
To determine and compare progression-free survival (PFS) in the experimental group and the control group by median time to progression in the respective arms | 6 months
To determine and compare overall survival (OS) in the experimental group and the control group | Until death
To analyse immunological activation by comparing patients with and without presence of tumour antigen recognizing CD8+ T cells | 6 months
To analyse clinical outcome by time to event endpoints (OS and PFS) | 6 months

CONTACTS AND LOCATIONS:
Locations (7):
- France (2):
  - Centre Georges-François Leclerc, Dijon
  - CHU de Rennes - Pontchaillou, Rennes
- Spain (5):
  - Hospital Universitario Quirón, Barcelona
  - Vall d'Hebron Univerity Hospital, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta - Institut Català d'Oncologia, Girona
  - Hospital 12 de octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid